CLINICAL TRIAL: NCT06604182
Title: Community-based HCV Testing and Treatment of People Who Inject Drugs: Innovate, Involve, Inspire
Brief Title: Innovate, Involve, Inspire
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Frontline AIDS (Other)
Collaborators: Alliance for the Public's Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERC.0004133
Record Dates: First submitted 2024-07-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HCV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HCV positive (Experimental): Eligible participants that are HCV infected.
  Interventions: Other: Community-based Simplified HCV Testing and Treatment Algorithm

INTERVENTIONS:
Other: Community-based Simplified HCV Testing and Treatment Algorithm — The distinctive features of CBSA are: (i) community-based service provision, substantially lowering the threshold for HCV services and eliminating the need to visit health care facilities for the majority of patients; (ii) the use of simple, once-daily, pan-genotypic HCV treatment regimens; (iii) a minimum of required laboratory tests and assessments; (iv) task sharing of essential functions from physicians to the case-managers; (v) integration of HCV testing and treatment with existing harm reduction services, addressing multiple health needs and facilitating patient-centered care.
  Other Names: CBSA

SUMMARY:
The study will test a Community-based Simplified HCV Testing and Treatment Algorithm (CBSA), implemented at community harm reduction fixed or mobile sites.

All potential participants with positive anti-HCV test will undergo diagnostic procedures including HCV-RNA testing. Those eligible for CBSA will be prescribed a fixed dose combination tablet: sofosbuvir/daclatasvir.

Sustained virologic response (SVR) will be assessed 12 weeks after treatment completion. All those who achieve SVR will be tested for HCV_RNA at six and 12 months after SVR12.

DETAILED DESCRIPTION:
People who inject drugs (PWID) bear the highest burden of the disease and due to multiple individual and structural barriers suffer from suboptimal access to accessing life-saving treatments. A range of interventions in the continuum of HCV testing and treatment have been suggested to address the specific needs of PWID. However, despite these advances, there is insufficient evidence on HCV integration in harm reduction from low-middle income countries, where the burden of HCV among people who inject drugs is the most significant.

This study seeks to contribute evidence to the global efforts in combating HCV among PWID, by identifying effective strategies to overcome barriers to testing and treatment, and ultimately advancing the goals of the WHO's global hepatitis strategy to eliminate HCV as a public health threat.

This is a mixed-methods observational cohort followed longitudinally with the core of the study intervention being the Community-Based Simplified HCV Testing and Treatment Algorithm (CBSA), described in detail below. CBSA is based on the latest WHO recommendations on HCV simplified service delivery, and clinical guidelines for non-specialized care settings. The distinctive features of CBSA are: (i) community-based service provision, substantially lowering the threshold for HCV services and eliminating the need to visit health care facilities for the majority of patients; (ii) the use of simple, once-daily, pan-genotypic HCV treatment regimens; (iii) a minimum of required laboratory tests and assessments; (iv) task sharing of essential functions from physicians to the case-managers; (v) integration of HCV testing and treatment with existing harm reduction services, addressing multiple health needs and facilitating patient-centered care. All potential participants with positive anti-HCV test will undergo diagnostic procedures including HCV-RNA testing. Those eligible for CBSA will be prescribed a fixed dose combination tablet: sofosbuvir/daclatasvir. Sustained virologic response (SVR) will be assessed 12 weeks after treatment completion. All those who achieve SVR will be tested for HCV_RNA at six and 12 months after SVR12.

The primary outcomes are based on the HCV treatment cascade: (a) Completing the pretreatment evaluation; (b) Initiating and completing the full DAA course; (c) Achieving SVR12; (d) Re-infection rate at six and 12 months after SVR12. Secondary outcomes include treatment motivation, adherence, quality of life, and treatment satisfaction. The qualitative component will explore client-level, provider-level, organizational, community-level, and structural factors influencing the integration of CBSA into harm reduction programs.

ELIGIBILITY:
Inclusion Criteria:

* Drug use in the past 90 days
* Age 18 and above
* Positive for HCV RNA

Exclusion Criteria:

* No meeting inclusion criteria
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1454 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants successfully completing HCV treatment | 15 months
  Hepatitis C screening, confirmation and treatment will be monitored for the number of confirmed positive participants that enroll and complete treatment. Suppression of the virus will be recorded per participant as well as re-infection rates up to 1 year after treatment was completed.

SECONDARY OUTCOMES:
The percentage of participants with treatment satisfaction using a tool called: Health seeking behavior and health service utilization | 15 months
  The tool will measure, in the last 6 months, the number of times participants 1. seeked medical assistance, 2. if assistance was provided, 3. the reason for not seeking assistance (if relevant) and 4. treatment satisfaction (if assistance was provided). These multiple measurements will be aggregated to give a score per participant used to classify participants into percentage with and without treatment satisfaction.

IPD SHARING:
Plan to Share IPD: No